CLINICAL TRIAL: NCT06362863
Title: A Randomized Controlled Study to Evaluate the Efficacy of Enteral Nutrition Biscuits in Inducing Remission in Moderate to Severe Crohn's Disease
Brief Title: Evaluation of Enteral Nutrition Biscuits for Inducing Remission in Moderate-to-severe Crohn's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ping An (Other)
Responsible Party: Sponsor-Investigator, Ping An, Professor, Renmin Hospital of Wuhan University
Organization: Renmin Hospital of Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2024-K027
Record Dates: First submitted 2024-03-24; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Crohn's Disease
Keywords: enteral nutrition; Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled study divided into intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral nutrition biscuits (Experimental): Addition of enteral nutritional biscuits to existing pharmacological treatment.
  Interventions: Dietary Supplement: enteral nutrition biscuits
- Conventional drug therapy (No Intervention): No nutritional intervention, use of existing medication.

INTERVENTIONS:
Dietary Supplement: enteral nutrition biscuits — Addition of enteral nutritional biscuits to existing pharmacological treatment.
  Arms: Enteral nutrition biscuits

SUMMARY:
By conducting a randomized controlled study of the role of enteral nutrition biscuits in the induction of remission in moderate-to-severe Crohn's disease, we will evaluate to investigate the role of enteral nutrition biscuits in the induction and remission phases of moderate-to-severe Crohn's disease; to assess patient adherence to enteral nutrition biscuits and the timing of their application; to assess the role of enteral nutrition biscuits in biologically refractory patients; and to assess the role of enteral nutrition biscuits in the remission of perianal, small bowel, and colonic lesions.

DETAILED DESCRIPTION:
This project is a randomized controlled study evaluating the effects of enteral nutrition biscuits during the induction and remission phases of moderate to severe Crohn's disease. The study subjects were patients with moderate to severe Crohn's disease, and the control group received conventional treatment with existing drugs; The experimental group added oral enteral nutrition biscuits to intervene on the basis of existing drugs. Evaluate the clinical response rates of patients at 2, 4, 8, 12, and 24 weeks after intervention; Nutritional status before and after intervention, incidence and severity of perianal lesions, and remission rate of small intestine and colon lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years old, gender is not limited
* Patients with a combination of clinical manifestations, laboratory examinations, endoscopy, imaging examinations and histopathological examinations to diagnose Crohn's disease for at least 6 months
* Patients with Crohn's disease with a CDAI score of > 220 and an HBI of ≥5
* Voluntarily signed written informed consent

Exclusion Criteria:

* Patients with newly diagnosed Crohn's disease, no history of treatment with 5-aminosalicylic acid, biological or immunological agents
* Current presence of an abscess or suspected abscess
* Positive results of stool culture or other intestinal pathogens
* Use of any antibiotics, prebiotics, probiotics, nutrition bars and enteral nutrition in the past 4 weeks
* Known hypersensitivity to any of the components administered in this study
* Severe infection (CTC AE> grade 2) within 4 weeks prior to the start of the study
* Patients who have recently undergone digestive surgery (< 1 month) or have not been completely cured
* Patients with severe gastrointestinal problems (such as life-threatening intestinal obstruction, perforation, and bleeding) requiring immediate treatment
* Have an underlying medical condition that affects treatment
* Pregnant or lactating women
* Positive for human immunodeficiency virus
* Known history of active pulmonary tuberculosis. Subjects with suspected active tuberculosis should be examined for chest x-ray, sputum, and exclusion by clinical signs and symptoms
* Patients with untreated chronic hepatitis B or hepatitis B virus carriers with chronic hepatitis B virus DNA exceeding 500 IU/mL, or patients with active hepatitis C should be excluded. Patients with inactive HBsAg, treated and stable hepatitis B patients (HBV DNA <500 IU/mL), and cured hepatitis C patients may be enrolled. Subjects with positive hepatitis C virus antibodies are eligible to participate in the study only if they have a negative HCV RNA test result
* Known history of psychotropic substance abuse, alcoholism, and drug abuse
* Any condition that, in the opinion of the investigator, the participant should be excluded from the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Crohn's disease activity index, CDAI | 2、4、8、12、24 weeks after intervention
  Assessment was performed using the Crohn's disease activity index (CDAI), with a clinical response defined as a CDAI score <150.

SECONDARY OUTCOMES:
Induced remission success rate | 2、4、8、12、24 weeks after intervention
  Probability of success of intervention in inducing CD remission.
Gastrointestinal Symptom Rating Scale (GSRS) score | 2、4、8、12、24 weeks after intervention
  Gastrointestinal Symptom Rating Scale (GSRS) score.
Gastrointestinal symptom remission | 4 weeks after intervention
  Gastrointestinal Symptom Rating Scale (GSRS) scores after 4 weeks of intervention.
Detection of antibody levels to the biologics used in sera from patients with secondary loss of response to the biologics | 1、4、8、12、24 weeks after intervention
  Detection of antibody levels to the biologics used in sera from patients with secondary loss of response to the biologics.
Incidence and severity of perianal lesions in both groups | 1、8、24 weeks after intervention
  Assess the incidence and severity of perianal lesions in both groups.
Rate of endoscopic remission of small bowel and colon lesions in both groups | 1、8、24 weeks after intervention
  Assess the rate of endoscopic remission of small bowel and colon lesions in both groups.
Changes in inflammatory biomarkers (C-reactive protein, fecal calreticulin) in both groups | 1、4、8、12、24 weeks after intervention
  Assess the changes in inflammatory biomarkers (C-reactive protein, fecal calreticulin) in both groups.
Adverse events and serious adverse events, safety and tolerability, with treatment-related adverse events and number of occurrences as assessed by CTCAE v5.0 | 1、4、8、12、24 weeks after intervention
  Adverse events and serious adverse events, safety and tolerability, with treatment-related adverse events and number of occurrences as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ping An, Principal Investigator — Renmin Hospital of Wuhan University

IPD SHARING:
Plan to Share IPD: No